CLINICAL TRIAL: NCT05313217
Title: The Influence of Spine Position on Measures of Lower Extremity Neural Sensitivity
Brief Title: Spine Position and Neural Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hartford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PRO20220124
Record Dates: First submitted 2022-03-28; First posted 2022-04-06 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Sciatic Nerve; Postural Lordosis; Nerve Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Intervention Model Description: Quasi-experimental single group laboratory study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neural tension testing (Experimental): All participants in this arm will undergo four tests: KEA, SLR, Slump, and Extended Slump
  Interventions: Diagnostic Test: Knee extension angle; Diagnostic Test: Straight Leg Raise; Diagnostic Test: Slump Test; Diagnostic Test: Extended slump test

INTERVENTIONS:
Diagnostic Test: Knee extension angle — Knee Extension Angle (KEA):
  * This test will be administered with an ankle-foot orthosis (AFO) maintaining the participants ankle in neutral.
  * The participant will lie supine on the examination table with the contralateral lower extremity (LE) stabilized on the support surface using a mobilization strap.
  * The hip of the lower being examined will be flexed to 90 degrees.
  * The participant will then actively straighten their lower leg while maintaining upper leg in same position
  * Once the participant feels they are at maximal knee extension (patient instructed to straighten leg as far as what is comfortable), the angle will be measured with iPhone Inclinometer.
  * Participant asked to report any symptoms they are feeling and where (recorded for qualitative analysis)
  Other Names: KEA
Diagnostic Test: Straight Leg Raise — Straight Leg Raise (SLR):
  * Position the participant in supine on the plinth with knees extended and L LE strapped to the plinth
  * The participant will keep the AFO donned on the R distal ankle to keep the ankle in neutral position.
  * A researcher will passively lift the participant's right leg moving at a slow but consistent pace of approximately 15 degrees per second, while keeping it straight until a significant resistance is detected or the participant reports a production of symptoms, whichever occurs first.
  * Measurement of the SLR angle will be assessed with iPhone inclinometer.
  * Participant asked to report any symptoms they are feeling and where (recorded for qualitative analysis)
  Other Names: SLR
Diagnostic Test: Slump Test — Slump Test Procedure:
  * Participant will be instructed to sit upright with their legs over the edge of table
  * AFO remains on R leg
  * Participant will sequentially flex trunk, look down at the floor
  * Participant will extend R knee until symptoms are felt. Measure of angle with iPhone inclinometer placed at superior aspect of medial malleolus
  * Participant asked to report any symptoms they are feeling and where (recorded for qualitative analysis)
Diagnostic Test: Extended slump test — Extended Slump Procedure:
  * Participant will be instructed to sit upright with their legs over the edge of table
  * AFO remains on R leg
  * Participant is asked to arch their lower back into maximal extension in sitting, stabilized to research bench to maintain hyper-lordosis posture.
  * The participant is asked first flex cervical spine, then to extend their knee until it reaches full ROM or symptoms are felt that limit ROM.
  * Knee extension ROM is assessed with iPhone inclinometer at superior aspect of medial malleolus.
  * Participant asked to report any symptoms they are feeling and where (recorded for qualitative analysis)

SUMMARY:
The purpose of this research study is to see if there is a relationship between the tightness of the hamstring muscles (muscles on the back of the thighs), reported sensations related to stretch of the nerves of the lower extremity, and different positions of participants' backs. We will investigate the qualitative differences as provided verbally by participants (sensation felt at maximum knee extension angle) and quantitative differences as provided by surface electromyographic (EMG) measurements of hamstring activity and inclinometer measures of the knee angle.

DETAILED DESCRIPTION:
The Slump Test, introduced by Maitland in 1978, has been a clinical staple for determining adverse neural tension or altered neurodynamics and neurosensitivity related to intradiscal derangement or stenotic narrowing of the lumbar spine. The slump test is a highly reliable, common clinical tool used to assess neural tissue mechanosensitivity in patients with both spinal and lower limb pain. However, it is unclear if the slump test can be used to differentiate between those with true adverse neural tension compared to those with neurosensitivity due to compression of the neuroforaminal interface. The positioning of the slump test places maximal tension on the neural tissues both caudally and cranially, either reducing knee extension angle (KEA) in the affected side as opposed to the unaffected side, provoking radicular symptoms, or both. Hall's research found that there was mechanical activity in the hamstring muscles that came on with neural tension testing. This finding can be used to objectively assess when a participant is at their peak tolerable limit of neural tension in specific trunk positions during the slump test. Observation and clinical experience suggest there may be a subset of individuals who have increased neural tension in the slump test during spinal extension (shortening of the nerves) as opposed to flexion (stretch of the nerves). To date, there has been little research that has objectively demonstrated how trunk position affects neural tension during the slump test. Our research aims to determine if there is a difference in patient reported symptoms and hamstring activity between trunk flexion and extension during the slump test with healthy, younger individuals with no recent history of low back pain (LBP) or related symptoms. We expect to find a difference in range of motion (ROM), symptoms, and hamstring activity when the slump test is done in spinal flexion as opposed to spinal extension. This research will help to establish the prevalence of greater sensitivity in the extended vs flexed posture and establish a normative set of symptoms as described by healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals between the ages of 18 and 65 without low back pain.

Exclusion Criteria:

* Known previous diagnoses of sciatica or disc herniation
* Diagnosis of scoliosis
* History of pain in the low back or back of the leg
* History of back surgeries
* Any recent hamstring injuries
* Any recent fractures
* History of osteoporosis
* Have feeling of pins and needles down the leg
* Have a known nervous system disorder
* Have a known systemic inflammatory condition
* Have Rheumatoid Arthritis
* Known history of cardiovascular issues
* Have a known connective tissue disorder
* Bowel/bladder issues
* Are or may be pregnant
* Type 1 or type 2 diabetes mellitus
* Active/history of cancer
* Allergy to adhesives
* Are actively involved in a lawsuit regarding personal bodily injury or receiving workman's compensation
* Currently taking/have recently taken antibiotics known as fluoroquinolones (ie. Cipro, Levaquin, Noroxin)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Knee Extension Angle | single testing session at enrollment
  A measurement of the degree of knee extension achieved during the KEA, Slump, and extended slump tests

SECONDARY OUTCOMES:
EMG activity, biceps femoris | single session at enrollment
  surface EMG activity of the biceps femoris during KEA, SLR, slump, and extended slump referenced to hamstring maximal voluntary isometric contraction
qualitative data- extent, nature, and intensity of pain | single testing session at enrollment
  for each test, the most distal extent of symptoms and intensity on the 11 point numeric pain rating scale will be collected. Participants will be asked to describe the nature of the symptoms experienced during the test (e.g. stretch, pain, pull, tingle, etc)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Swanson, PT, DSc, Principal Investigator — University of Hartford
Locations (1):
- University of Hartford, West Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon request following completion of this study
Supporting Information: Study Protocol, SAP
Time Frame: Following study completion and manuscript submission
Access Criteria: upon request

REFERENCES:
- [Derived] Swanson B, McCarthy J, Clark E, Norman O, Wilson O. The influence of spine position on measures of lower extremity neural sensitivity. J Back Musculoskelet Rehabil. 2025 Aug 21:10538127251370575. doi: 10.1177/10538127251370575. Online ahead of print. PMID 40836858